CLINICAL TRIAL: NCT03101254
Title: A Phase I/II Study of LY3022855 With BRAF/MEK Inhibition in Patients With Melanoma
Brief Title: LY3022855 With BRAF/MEK Inhibition in Patients With Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Elizabeth Buchbinder, MD, Elizabeth Buchbinder MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-030
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — LY3022855; Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib (Experimental): * Starting dose level of LY3022855 50mg IV administered intravenously every week
  * Vemurafenib 960 mg BID administered by mouth twice daily
  * Cobimetinib 60 mg administered by mouth once daily on days 1-21of each cycle
  Interventions: Drug: LY3022855; Drug: Vemurafenib; Drug: Cobimetinib
- Phase I: Dose Level 2: LY3022855 (75mg) + Vemurafenib + Cobimetinib (Experimental): * LY3022855 50mg IV administered intravenously every week
  * Vemurafenib 960 mg BID administered by mouth twice daily
  * Cobimetinib 60 mg administered by mouth once daily on days 1-21of each cycle
  Interventions: Drug: LY3022855; Drug: Vemurafenib; Drug: Cobimetinib
- Phase I: Dose Level 3: LY3022855 (100mg) + Vemurafenib + Cobimetinib (Experimental): * LY3022855 100mg IV administered intravenously every week
  * Vemurafenib 960 mg BID administered by mouth twice daily
  * Cobimetinib 60 mg administered by mouth once daily on days 1-21of each cycle
  Interventions: Drug: LY3022855; Drug: Vemurafenib; Drug: Cobimetinib
- Phase II: LY3022855 (MTD) + Vemurafenib + Cobimetinib (Experimental): * MTD of LY3022855 was not established
  * Vemurafenib planned 960 mg BID administered by mouth twice daily
  * Cobimetinib planned 60 mg administered by mouth once daily on days 1-21of each cycle
  Interventions: Drug: LY3022855; Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: LY3022855 — LY3022855 is a colony-stimulating factor-1 receptor (CSF-1R) inhibitor
Drug: Vemurafenib — Vemurafenib is a BRAF inhibitor that works by blocking altered BRAF proteins from stimulating the growth of melanoma cancer cells
  Other Names: Zelboraf
Drug: Cobimetinib — Cobimetinib works by blocking a protein called MEK that has been known to promote melanoma growth
  Other Names: Cotellic

SUMMARY:
This research study is studying a combination of targeted therapies as a possible treatment for advanced melanoma that was found to have a BRAF V600E or BRAF V600K genetic mutation

The interventions involved in this study are:

* LY3022855
* Vemurafenib
* Cobimetinib

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved LY3022855 as a treatment for any disease.

The FDA has approved vemurafenib and cobimetinib as treatment options for this disease.

LY3022855 is a colony-stimulating factor-1 receptor (CSF-1R) inhibitor. It is a human monoclonal antibody. A monoclonal antibody is a type of protein made in the laboratory that can locate and bind to substances in the body, including tumor cells. By binding to the tumor cells, the antibody might prevent the tumor cell from growing and spreading. LY3022855 is being developed as a treatment for patients with advanced cancer.

Vemurafenib and cobimetinib attack different proteins that promote the growth of cancerous cells. Vemurafenib is a BRAF inhibitor that works by blocking altered BRAF proteins from stimulating the growth of melanoma cancer cells. Cobimetinib works by blocking a protein called MEK that has been known to promote melanoma growth. In order to participate in the study, participant's disease needs to be tested positive for a mutation (a permanent change in the DNA sequence of a gene) of the BRAF gene that belongs to a class of genes known as oncogenes. When mutated, oncogenes have the potential to cause normal cells to become cancerous. Once the BRAF gene is mutated, the normal functioning of the BRAF protein may be changed.

In this research study, the investigators are combining LY3022855 with vemurafenib and cobimetinib in the hopes that the LY3022855 will enhance how your cancer responds to vemurafenib and cobimetinib.

ELIGIBILITY:
Inclusion Criteria:

* For enrollment to the phase I portion: participants must have a histologically confirmed melanoma with a BRAF V600E or BRAF V600K mutation (identified via NextGen sequencing using the DFCI/BWH OncoPanel or any CLIA-certified method) that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective.
* For enrollment to the phase II portion: participants must have a histologically confirmed melanoma with a BRAF V600E or BRAF V600K mutation (identified via NextGen sequencing using the DFCI/BWH OncoPanel or any CLIA-certified method) and cannot have received prior BRAF or MEK inhibitor therapy.
* Participants enrolling to the phase I portion of the trial must have evaluable or measurable disease (see Section 11 for definitions).
* Participants enrolling to the phase II portion of the trial must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Age ≥ 18 years. As no dosing or adverse event data are currently available in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* ECOG performance status 0 - 1 (see APPENDIX A).
* Participants must have normal organ and marrow function as defined below:
* Absolute neutrophil count ≥ 1.5 K/uL
* Platelets ≥ 100 K/uL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN
* Serum creatinine ≤ 1.5 × institutional ULN
* PT-INR ≤ 1.5 × institutional ULN (for participants on anticoagulation therapy, ≤ 1.5 × their baseline value)
* aPTT ≤ 1.5 × institutional ULN (for participants on anticoagulation therapy, ≤ 1.5 × their baseline value)
* Participants must have a left ventricular ejection fraction (LVEF) ≥ 50%.
* Participants must have a QTc of ≤ 470 msec on the screening EKG.
* The effects of LY3022855 on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of LY3022855 administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must have archival tumor tissue available. Participants without archival tissue may be enrolled at the discretion of the principal investigator.

Exclusion Criteria:

* Participants who have had chemotherapy, radiotherapy, biologic therapy, major surgery, or another investigational agent within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Participants who have not recovered to ≤ CTCAE grade 1 or baseline from toxicity as a result of previous cancer treatment prior to entering the study (with the exception of alopecia and peripheral neuropathy which can be ≤ grade 2).
* For enrollment to the phase II portion: participants who have received prior BRAF or MEK inhibitor therapy.
* Participants with known untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with a history of brain metastases that have been treated, are no longer taking corticosteroids, and have been stable on imaging for ≥ 4 weeks following the last date of treatment are permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LY3022855, vemurafenib, or cobimetinib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because LY3022855 is an anti-cancer agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LY3022855, breastfeeding should be discontinued if the mother is treated with LY3022855. These potential risks may also apply to the other agents used in this study.
* Participants with a known history of HIV are ineligible because of the potential for pharmacokinetic interactions with LY3022855, vemurafenib, and cobimetinib with antiretroviral agents. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Participants with a personal or family history of long QT syndrome.
* Participants with a history of a second primary malignancy. Exceptions include: patients with a history of malignancies that were treated curatively and have not recurred within 3 years prior to study entry; resected basal and squamous cell carcinomas of the skin, and completely resected carcinoma in situ of any type.
* Participants with impairment of GI function or GI disease that may significantly alter the absorption of vemurafenib and cobimetinib in the opinion of the treating investigator (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Participants who are unable to swallow or retain oral medication.
* Participants that require co-administration of strong or moderate CYP3A inhibitors, as these medications may alter vemurafenib and cobimetinib concentrations.
* Participants who require treatment with medications that are strong or moderate CYP3A inducers, as these medications may alter the concentration of cobimetinib.
* Participants with evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Buchbinder, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrolled from June 2017 to March 2019.
Groups:
- Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib: * LY3022855 50mg IV administered intravenously every week
  * Vemurafenib 960 mg BID administered by mouth twice daily
  * Cobimetinib 60 mg administered by mouth once daily on days 1-21of each cycle
- Phase I: Dose Level 2: LY3022855 (75mg) + Vemurafenib + Cobimetinib: * LY3022855 75mg IV administered intravenously every week
  * Vemurafenib 960 mg BID administered by mouth twice daily
  * Cobimetinib 60 mg administered by mouth once daily on days 1-21of each cycle
Period: Overall Study
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib | Phase I: Dose Level 2: LY3022855 (75mg) + Vemurafenib + Cobimetinib | Phase I: Dose Level 3: LY3022855 (100mg) + Vemurafenib + Cobimetinib | Phase II: LY3022855 (MTD) + Vemurafenib + Cobimetinib
Started | 5 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I]
Description: DLT is based on CTCAE v4.03. DLT refers to toxicities experienced during the first cycle of treatment that are possibly, probably, or definitely related to the study medication regimen, and grade or category outlined in protocol section 5.4.
Time Frame: Participants were assessed cycle 1 on day 1, 8, 15 and 22. The observation period for DLT evaluation was the first cycle (28 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib
Number analyzed (Participants) | 5
Participants | 1

2. Primary Outcome: LY3022855 Maximum Tolerated Dose (MTD) With Vemurafenib and Cobimetinib Combination [Phase I]
Description: See previous primary outcome measure for the DLT defination. A conventional algorithm (3+3 design) will be used to identify the MTD, escalating on 0/3 or 1/6 DLTs, and de-escalating if two DLTs are encountered. The MTD will be the highest dose level at which ≤ 1/6 subjects experience a DLT. If dose level 1 is discovered to be intolerable (with 2/3 or ≥ 2/6 subjects experiencing a DLT), the trial will be discontinued.
Time Frame: Participants were assessed cycle 1 on day 1, 8, 15 and 22. The observation period is the first cycle (28 days).
Measure: Number; unit: mg
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib
Number analyzed (Participants) | 5
mg | 50

3. Secondary Outcome: Median Progression-Free Survival (PFS) [Phase I]
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria.
Time Frame: Disease was assessed radiologically at baseline and after treatment every 3-4 months. Median follow-up for survival was 202 days with maximum of 480 days.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib
Number analyzed (Participants) | 5
months | 3.7 [1.9 to 37.2]

4. Secondary Outcome: Overall Response Rate (ORR) [Phase I]
Description: The overall response rate (ORR) was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria.
Time Frame: Radiologic measurements is performed at Cycle 2 Day 28 and at the day 28 of every 2 cycles of treatment thereafter. Median treatment duration is 112 days (range 56 - 1008 days ).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib
Number analyzed (Participants) | 5
percentage of participants | 20.0 [1 to 66]

5. Secondary Outcome: Grade 3-5 Treatment-related Toxicity Rate [Phase II]
Description: All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4.03 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.
Time Frame: AE evaluated on treatment on each cycle at day 1, 8, 15 and 22. Median treatment duration for this study cohort was 112 days (range 56 - 1008 days).
Population: Phase II never started
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Measured while on-treatment of 1 cycle = 28 days. Mortality observation period is median of 202 days and maximum of 480 days.
Description: A serious adverse event (SAE) is any adverse event during this study that results in one of the following outcomes: death; hospitalization for greater than 24 hours; prolonging an existing inpatient hospitalization; a life-threatening experience (that is, immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; considered significant by the investigator for any other reason. All others are classified as other adverse event (OAE).
Arm/Group | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib (N=5)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Gallbladder infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1: LY3022855 (50mg) + Vemurafenib + Cobimetinib (N=5)
Anemia (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 3
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 2
Skin infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Cholesterol high (Investigations) | 1
CPK increased (Investigations) | 2
Creatinine increased (Investigations) | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT03101254/Prot_SAP_000.pdf